CLINICAL TRIAL: NCT04744311
Title: Translation and Validation of the Turkish Version of the Obstetric QoR-11 Questionnaire for the Evaluation of Recovery After Caesarean Section: the ObsQoR-11T Questionnaire
Brief Title: Translation and Validation of the Turkish Version of the ObsQoR-11 Questionnaire
Acronym: ObsQoR-11T
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Umut Kara, Consultant, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Other Study IDs: 2020-506
Record Dates: First submitted 2021-02-01; First posted 2021-02-08 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Patient Reported Outcome Measures; Quality of Recovery; Cesarean Section; General Anesthesia
Keywords: Questionnaire Obstetric Quality-of-recovery 11 (ObsQoR-11T)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ObsQoR-11T Questionnaire — The ObsQoR-11T questionnaire consists of 11 items assessing different aspects of postpartum recovery: physical comfort and pain, physical independence and emotional status. If the patient is not able to read the questionnaire herself, a third person can ask the questions orally to the patient. Each item is scored from 0 to 10 and the total score is the sum of the score for each item, which is a score from 0 to 110.

SUMMARY:
Ciechanowicz et al. developed and validated a postpartum recovery score for women with a caesarean section: the ObsQoR-11. The psychometric validation of the ObsQoR-11 confirms its reliability, its response to change, its acceptability and its feasibility. The use of this score allows the investigators to quantify the quality of the patient's recovery between 0 and 110, by allocating a score from 0 to 10 for each item. ObsQoR-11 has not yet been validated for use in Turkish. Therefore the investigators aimed to psychometrically evaluate the Turkish translated version of the ObsQoR-11 in a Turkish cohort of women.

DETAILED DESCRIPTION:
Recovery after caesarean section is a complex process, depending on the characteristics of the patient and the anaesthesia. Scales for measuring the quality of post-operative recovery have been developed. Ciechanowicz et al. developed and validated a postpartum recovery score for women with a caesarean section: the ObsQoR-11. This multidimensional scale is a questionnaire of 11 items evaluating: moderate pain, severe pain, nausea and vomiting, feeling of discomfort, shivering, feeling of comfort, ability to mobilize, ability to carry the newborn, ability to feed, ability to groom alone, and finally feeling of self-control. The investigators aimed to validate the translated version of the Turkish ObsQoR-11 scale.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old)
* Turkish-speaking
* Admitted for cesarean section
* Able to answer the questionnaire, alone or with the help of a third party
* Agreeing to participate in the study

Exclusion Criteria:

* Psychiatric or neurological pathology

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted for cesarean section
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Validity of ObsQoR-11T questionnaire | At 24 hours after caesarean section
  Evaluate the validity of the Turkish version of the ObsQoR-11 to assess postoperative recovery

CONTACTS AND LOCATIONS:
Locations (1):
- SBÜ Gülhane Education and Training Hospital, Etlik, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ciechanowicz S, Setty T, Robson E, Sathasivam C, Chazapis M, Dick J, Carvalho B, Sultan P. Development and evaluation of an obstetric quality-of-recovery score (ObsQoR-11) after elective Caesarean delivery. Br J Anaesth. 2019 Jan;122(1):69-78. doi: 10.1016/j.bja.2018.06.011. Epub 2018 Jul 31. PMID 30579408
- [Background] Ciechanowicz S, Howle R, Heppolette C, Nakhjavani B, Carvalho B, Sultan P. Evaluation of the Obstetric Quality-of-Recovery score (ObsQoR-11) following non-elective caesarean delivery. Int J Obstet Anesth. 2019 Aug;39:51-59. doi: 10.1016/j.ijoa.2019.01.010. Epub 2019 Feb 2. PMID 30885691